CLINICAL TRIAL: NCT03748290
Title: The Effect of Preventional Drug Therapy on Pain Regulation Mechanisms Among Spinal Cord Injury Patients Who Have Yet to Develop Central Pain
Brief Title: Effect of Preventional Drug Therapy on Pain Regulation Mechanisms Among SCI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Gabriel Zeilig, Director of the Neurological Rehabilitation Department, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4686-17-SMC
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Spinal Cord Injuries; Central Pain Syndrome
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The placebo pills will be purchased from Trilog, which is licensed and licensed by the Ministry of Health to prepare random drug kits (the company has an agreement with Sheba). The drug will be used by the company that supplies the drug and placebo, so that the researchers in the study did not know which treatment was given to each patient. This information will be received at the end of the study, or if the subjects for any reason participate in the research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- People with a SCI who will receive Lyrica 75mg for 12 weeks (Experimental)
  Interventions: Drug: Pregabalin
- People with a SCI who will receive Placebo for 12 weeks (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 75 mg for 12 weeks
  Other Names: Lyrica
  Arms: People with a SCI who will receive Lyrica 75mg for 12 weeks
Drug: Placebo Oral Tablet — Placebo Oral Tablet
  Arms: People with a SCI who will receive Placebo for 12 weeks

SUMMARY:
Central neuropathic pain (CNP) is defined as chronic pain due to injury or disease in the central nervous system. This pain is most common among people with a spinal cord injuries (SCI), with a prevalence of about 50%. The central pain usually develops within a few months of spinal cord injury - and this period is significance in terms of this research work. This pain is one of the most complex and challenging pain syndromes. One of the reasons for this stems from its adherence to most treatments. Another reason is that there is partial information about the mechanism responsible for its development. Animal studies suggest that it is possible to prevent and / or reduce its development or reduce its strength by preventive treatment (given immediately after the injury). Currently, the treatments found to prevent or reduce central pain in animals are anti Inflammation and neuronal excitability suppressors such as interleukin 10.

The purpose of this study,is to explore whether pre-treatment with pregabalin prior to the development of the central pain will prevent the incidence of pain or reduce its intensity by improving pain regulation and reducing hypersensitivity.

The goal of the pharmacotherapy is to reduce the hypersensitivity- lyrica is used to reduce chronic neuropathic pain by reducing the degree of hypersensitivity in the pain system.

the objectives of this study are to examine whether early treatment of central pain can prevent or reduce the incidence of pain by improving pain regulation and reducing hypersensitivity. That is, whether there will be a difference between those who take Lyrica-Pregabalin (a drug that reduces hypersensitivity of pain) compared to placebo.

Methods: A randomized, double-blind, placebo-controlled study in which people with a fresh SCI will receive lyrica or placebo as soon as possible from their arrival at the rehabilitation hospital for 2-3 months during which pain system characteristics will be measured and monitored for central pain development.

ELIGIBILITY:
Inclusion Criteria:

* People with a Spinal injury below C3 2-3 weeks after the injury
* Cognitive, mental, and verbal state (understanding and speech) that allows for voluntary cooperation in research and compliance with instructions

Exclusion Criteria:

* Pregnant women
* Other neurological diseases (such as head trauma)
* Other systemic diseases that affect the sensation (such as uncontrolled diabetes).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Central Pain: monitored for any complaints | 12 weeks
  Subjects will be constantly monitored for any complaints of pain and the pain will be diagnosed. Upon a diagnosis of central neuropathic pain, the first outcome is achieved
Central neuropathic pain severity: McGill pain questionnaire | 12 weeks
  Two major quantitative parameters are derived: (1) the number of words chosen (NWC) by the subject from a list of descriptors (total score ranges between 0-19), and (2) the pain rating index (PRI)- based on summing the rank values of these words (total score ranges between 0-65). Higher values represent worse outcome.
Pain modulation capacity - Visual analog scale (VAS) | 12 weeks
  0=no pain, 10=most intense pain imaginable, Higher values in the VAS represent worse outcome. This outcome will be assessed with the conditioned pain modulation and the temporal summation experimental paradigms.
  The Conditioned Pain Modulation (CPM) paradigm is an experimental paradigm the results of which indicate on the capacity of the pain modulation systems. The magnitude of CPM will be the outcome measure and it is calculated by subtracting a pain rating on the VAS of a noxious stimulus administered alone and in the presence of another, remote stimulus.
  The temporal summation of pain (TSP) paradigm is an experimental paradigm the results of which indicate on the level of excitability of the pain system. The magnitude of TSP will be the outcome measure and it is calculated by subtracting a pain rating on the VAS given at the termination of a continuous noxious stimulus from that given at the beginning of the same stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Gabi Zeilig, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center rehabilitaion facility, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided